CLINICAL TRIAL: NCT06000410
Title: A Phase 3 Prospective, Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy of Amniotic Suspension Allograft (ASA) in Patients With Osteoarthritis of the Knee
Brief Title: A Study to Evaluate the Efficacy of Amniotic Suspension Allograft in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22 OA 003 ASA
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Arthritis; Joint Disease; Musculoskeletal Diseases; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized, double-blind, placebo-controlled study of ASA in patients with OA of the knee. Patients will be randomly assigned in a 1:1 ratio to receive a single IA injection of 2 mL of ASA (plus 2 mL of normal saline) or 4 mL of normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) All clinic staff who may be involved in making assessments of safety will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASA (Experimental): Participants receive a single IA injection of 2 mL of ASA (plus 2 mL of normal saline)
  Interventions: Biological: Amniotic Suspension Allograft
- Placebo (Placebo Comparator): Participants receive a single IA injection of 4 mL of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Amniotic Suspension Allograft — This investigational product is a cryopreserved product derived from human amnion and cells from the amniotic fluid.
  Arms: ASA
Drug: Placebo — Matching placebo is 0.9% normal saline: 4 mL to be injected IA.
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of ASA compared to placebo in the management of osteoarthritis (OA) symptoms of the knee.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled Phase 3 study of ASA in patients with OA of the knee. Initially, 474 subjects are planned for inclusion in this study using a group sequential design with an interim analyses and a final analysis. Patients will be randomly assigned in a 1:1 ratio to receive a single intra-articular (IA) injection of 2 mL of ASA (plus 2 mL of normal saline) or 4 mL of normal saline on Day 1.

They will have serial assessments of knee pain, function, and symptoms scores, as well as safety assessments for up to 52 weeks after administration of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older
* Diagnosis of OA of the index knee by a combination of clinical and radiographic findings.
* OA of the index knee with Kellgren and Lawrence radiographic classification (Grades 2-4 inclusive),
* Patients who have failed to adequately respond for at least 6 months to at least two osteoarthritis therapies within the last 12 months
* Overall index knee pain score above minimum required WOMAC Pain scale.
* Body mass index < 40 kg/m2
* Using birth control, sterile or post-menopausal.
* Able to understand and provide written informed consent

Exclusion Criteria:

* Kellgren and Lawrence radiographic grade 1 OA of the knee
* Use of pain medication less than 5 days before the baseline visit
* Regular use of anticoagulants
* Symptoms that could indicate meniscal displacement or an IA loose body.
* Corticosteroid injection into the index knee within 3 months prior to screening.
* Viscosupplement or any other autologous or allogeneic product into the index knee within 6 months prior to screening.
* Patients with known hypersensitivity reactions to ASA or any of its constituents.
* Knee surgery on the index knee within 12 months prior to screening and/or planned knee surgery during the study
* Knee surgery on the contralateral knee within 6 months prior to screening and/or planned knee surgery during the study
* Acute index knee trauma within 3 months prior to screening
* Knee effusion requiring aspiration of the index or contralateral knee within 3 months prior to screening.
* Contralateral knee pain above limits defined in the protocol
* Current therapy with any immunosuppressive therapy or medical conditions likely to require systemic steroids during the study.
* Any active or systemic infection including infection of the index knee joint or breakdown or disease of the index knee skin/soft tissues.
* Clinically significant intercurrent illness, medical condition, non-knee pain, or medical history that would jeopardize patient safety, limit participation, or compromise interpretation of data derived from the patient
* Active alcohol or substance use disorder, or any other reason that would make it unlikely that the patient will comply with study procedures
* Females who are pregnant or lactating
* Participation in another clinical trial within the 30 days (or 5 half-lives of the investigational compound, whichever is longer) before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
The difference in change from baseline in WOMAC Pain scale at 6 months between ASA- and placebo-treated patients | Baseline to Week 26
  The WOMAC is widely used in the evaluation of hip and knee OA. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain, stiffness, and physical function. The WOMAC measure has been used in clinical trials to evaluate the efficacy of surgical treatments, medicinal and biological products, devices, and physical therapies.

SECONDARY OUTCOMES:
The difference between changes from baseline for ASA- and placebo- treated patients in WOMAC Function at 6 months | Baseline to Week 26
  The WOMAC is widely used in the evaluation of hip and knee OA. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain, stiffness, and physical function. The WOMAC measure has been used in clinical trials to evaluate the efficacy of surgical treatments, medicinal and biological products, devices, and physical therapies.
The difference between changes from baseline for ASA- and placebo-treated patients in the OMERACT-OARSI responder rate at 6 months | Baseline to Week 26
  The OMERACT-OARSI core domain set for clinical trials in hip and/or knee osteoarthritis responder criteria will be used to assess whether a patient is a responder or not.
The difference between changes from baseline for ASA- and placebo-treated patients in WOMAC Pain at 3 months | Baseline to Week 12
  The WOMAC is widely used in the evaluation of hip and knee OA. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain, stiffness, and physical function. The WOMAC measure has been used in clinical trials to evaluate the efficacy of surgical treatments, medicinal and biological products, devices, and physical therapies.

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Fiel Family & Sports Medicine, Tempe, Arizona
  - Horizon Clinical Research, La Mesa, California
  - Neurovations Research, Napa, California
  - Infinity Clinical Research, Norco, California
  - Dream Team Clinical Research, Pomona, California
  - Stanford Medicine, Redwood City, California
  - TriWest Research Associates, San Diego, California
  - AppleMed Research Group, LLC., Miami, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - CenExcel/ACMR, Atlanta, Georgia
  - Vista Clinical Research, Newnan, Georgia
  - Chicago Clinical Research Institute Inc., Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Advanced Quality Medical Research, Inc, Orland Park, Illinois
  - MediSphere Medical Research Center, Evansville, Indiana
  - Sinai Hospital, Baltimore, Maryland
  - Klein & Associates M.D., P.A., Hagerstown, Maryland
  - Skylight Health Research, Burlington, Massachusetts
  - Oakland Medical Research, Troy, Michigan
  - Sundance Clinical Research, St Louis, Missouri
  - Physician Research Collaboriation, LLC, Lincoln, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Northwell Health, New York, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - West Clinical Research, Morehead City, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Tekton Research, Austin, Texas
  - Cedar Health Research, LLC, Burleson, Texas
  - ClinRXResearch INC, Carrollton, Texas
  - Zenos Clinical Research, Dallas, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - Spectrum Medical, Inc., Danville, Virginia
  - Spokane Joint Replacement Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No